CLINICAL TRIAL: NCT06323343
Title: Mobile Video Education to Improve Patient Clinician Communication During Prenatal Clinic Visits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Mir A Basir, Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 00040976
Record Dates: First submitted 2024-03-14; First posted 2024-03-21 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Patient Empowerment
Keywords: Prenatal care; Congenital abnormalities; Communication; Mobile health
MeSH Terms: conditions — Patient Participation; Congenital Abnormalities; Communication

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Video Intervention (Experimental): Participants assigned to the video intervention group receive a text message prior to their prenatal fetal anomaly appointment. Embedded in that text message is a link to an animated video which provides education on best practices of communicating with providers.
  Interventions: Other: Video Intervention
- Webpage links (Active Comparator): Participants assigned to the webpage links group receive links to the clinic's publicly available webpages prior to their prenatal fetal anomaly appointment. The webpages provide background about the providers and services available as well as a tour of the clinic.
  Interventions: Other: Webpage links

INTERVENTIONS:
Other: Video Intervention — Animated video delivered by text message to prepare parents to communicate with physicians at their upcoming appointment for a fetal anomaly concern.
  Arms: Video Intervention
Other: Webpage links — Links to publicly available webpages about the fetal concerns clinic where the participants' appointments are scheduled.
  Arms: Webpage links

SUMMARY:
The goal of this clinical trial is to test an animated video delivered by text message in patients whose pregnancies are complicated with fetal anomalies. The main question it aims to answer is: Does the video intervention prepare parents to talk to the doctors during prenatal appointments?

Participants will be randomized to receive either the video intervention or links to the clinic's webpages. They will complete an enrollment survey before their appointment and a follow up survey after their appointment.

The researchers will compare the video and webpage groups to see which group reports engaging in more of the identified best-practices of communication.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patient scheduled for an appointment at the Children's Wisconsin Fetal Concerns Center for a fetal anomaly.
* Able to speak and understand English (intervention videos are only currently available in English).
* Age of 18 years or older.

Exclusion Criteria:

* Pregnant patient's appointment at Children's Wisconsin Fetal Concerns center is not for a fetal anomaly (e.g., screening only, past pregnancy with anomaly only cause of appointment)
* Pregnant patient is considering termination of pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-06-15 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Parents' communication behaviors measure | Administered 1 day after appointment
  Participants' self-reported behaviors during the prenatal fetal anomaly appointment, on a scale from 0-14, with higher scores indicating a higher rate of best-practice communication behaviors.

CONTACTS AND LOCATIONS:
Locations (1):
- Fetal Concerns Center Children's Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No